CLINICAL TRIAL: NCT06464588
Title: A Phase 1 Open-Label Study of the Safety of Intravenous Allogeneic Neonatal Mesenchymal Cells (nMSCs) in Young Adult (1A) and Pediatric (1B) Patients With Dilated Cardiomyopathy (DCM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Principal Investigator, William T. Mahle, Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004268
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Dilated Cardiomyopathy
Keywords: Dilated Cardiomyopathy; Neonatal Mesenchymal Cells (nMSCs)
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adult Cohort (Experimental): Adults (18-30 years) will be enrolled into all dose levels (as tolerated) of Phase 1A. Open label nMSCs will be administered intravenously in the following defined dose groups. The rate of infusion will be approximately 30- 60 minutes at 0, 15 and 30 days, with escalating dose levels:
  * Dose level 1: 5.0x107 nMSCs at 0, 15 and 30 days
  * Dose level 2: 1.0.x108 nMSCs at 0, 15 and 30 days
  * Dose level 3: 2.5x108 nMSCs at 0, 15 and 30 days
  Dose escalation will follow 3+3 study design parameters. The next dosing group will be initiated at least one month after the last subject in a particular dose level has received the last dose treatment. Once MTD has been determined, 3 additional patients will be enrolled to ensure a total of 6 patients are enrolled in MTD level for confirmation.
  Interventions: Biological: Allogeneic Neonatal mesenchymal stromal cells (nMSCs)
- Pediatric Cohort (Experimental): Pediatric participants (ages 4 years-18 years) will be enrolled into dose level as determined in Phase 1B (3+3 study design; open label).
  nMSCs will be administered intravenously in the following defined dose groups. The rate of infusion will be approximately 30- 60 minutes at 0, 15 and 30 days, with escalating dose levels:
  * Dose Level 1: 0.7x106 nMSCs/kg
  * Dose Level 2: 1.43x106 nMSCs/kg
  * Dose Level 3: 2.85x106 nMSCs/kg
  Dose escalation will follow 3+3 study design parameters. The next dosing group will be initiated at least one month after the last subject in a particular dose level has received the last dose treatment. Once MTD has been determined, 3 additional patients will be enrolled to ensure a total of 6 patients are enrolled in MTD level for confirmation.
  Following intravenous delivery of nMSCs, patients will be followed at 3 months, 6 months and 1 year from the last infusion to complete all safety and efficacy assessments.
  Interventions: Biological: Allogeneic Neonatal mesenchymal stromal cells (nMSCs)

INTERVENTIONS:
Biological: Allogeneic Neonatal mesenchymal stromal cells (nMSCs) — nMSCs will be administered intravenously in the predefined dose per each group. The rate of infusion will be approximately 30- 60 minutes at 0, 15 and 30 days, with escalating dose levels.
  Other Names: nMSCs infusions

SUMMARY:
This is a Phase 1 study to determine the safety and efficacy of allogeneic neonatal mesenchymal stromal cells (nMSCs) for the treatment of Dilated Cardiomyopathy. The purpose of the study is to help doctors and scientists learn if allogeneic neonatal mesenchymal stromal cells (nMSCs) infusions are a safe and effective way to improve cardiac function and left ventricular ejection fraction.

DETAILED DESCRIPTION:
This study is a single site open label study with 2 phases. The 2 phases will be broken into an adult group Phase 1A with group pediatric group Phase 1B. This study will enroll patients between the ages of 4 years and 30 years old. The investigators will be looking at the safety, feasibility, and maximum tolerated dose of allogeneic neonatal mesenchymal stromal cells (nMSCs) as defined by freedom from CTCAE or Grade 3 AE that is probably or definitely related to the IP throughout the duration of the study.

A minimum of 9 and a maximum of 18 patients will be enrolled into both Phase 1A adult groups and 1B pediatric groups. Phase 1A subjects will receive study products with doses defined by the study group and Phase 1B will begin after all adult subjects have completed Phase 1A infusions, FDA and a DSMC review. All pediatric subjects will receive study product dosed per body weight in the defined study group.

Allogeneic neonatal mesenchymal stromal cells (nMSCs) will be infused via IV every 30 days for a total of 3 infusions. A check-in will be scheduled the morning after each infusion for pediatric patients. There will be a baseline visit before allogeneic neonatal mesenchymal stromal cells (nMSCs) therapy is initiated, followed by a phone call 30 days after the last infusion. There will be in person visits at 3-month, 6 months, and 1 year mark. The total duration for each patient will be 14 months.

Labs will be collected at baseline, during nMSC infusions, and at in person follow up visits to assess cardiac function. Any leftover blood samples may be stored for future research by the sponsor of the study. Echocardiograms will be completed at baseline, and 3 month-, 6 month-, and 1-year visits to look at left ventricular ejection fraction and electrocardiograms will be completed to provide measures of cardiac rhythm or rhythm. Other assessments include physical exam, 6-minute walk test, Cardiac MRI, vital signs, PedsQL questionnaire for pediatrics and The Kansas City Cardiomyopathy Questionnaire for adults.

It is expected to recruit 18-36 participants through face-to-face encounters between participants and study staff during clinical encounters at Children's Healthcare of Atlanta and Emory Health care system, Clinicaltrials.gov registration, and Institutional Review Board approved advertisements to surrounding hospitals with cardiac programs. Patients will also be recruited through MyChart. If identified as eligible to participate, the study team will seek approval by the subjects' primary cardiologist and consent and/or assent with the permission of the parent or legally authorized representative, will occur in person during a baseline visit.

After allogeneic neonatal mesenchymal stromal cells (nMSCs) infusions, pediatric patients will be provided an overnight stay at Ronald McDonald House, or a hospital affiliated hotel in case of any unanticipated effects and follow up visits the next morning. This is so pediatric patients are near the hospital for such events. Adults will not be required to stay overnight for a follow-up visit. There will be financial compensation for each study visit, and patients will be reimbursed for parking.

ELIGIBILITY:
Inclusion Criteria

* Phase 1A: Age greater than or equal to 18 years and less than 30 years (≥18 years, <30 years).
* Phase 1B: Age greater than or equal to 4 years and less than 18 years (≥4 years, <18 years)
* Subjects must be able to sign their own consent for Phase 1A of the study.
* Diagnosis of dilated cardiomyopathy (DCM) defined as

  * Any Congenital Cardiac Malformation with systemic ventricular systolic dysfunction; Idiopathic Cardiomyopathy; Familial/Inherited and/or Genetic Cardiomyopathy; History of Myocarditis; Acquired (Chemotherapy, Iatrogenic, Infection, Rheumatic, Nutritional); Ischemic (e.g. Kawasaki Disease, post-operative); Left ventricular noncompaction; Coronary Artery Disease
  * Left ventricular ejection fraction less than or equal to 45% documented by two-dimensional echocardiogram or cardiac MRI within the prior six months.
  * Left ventricular dilation as defined by echocardiography left ventricular and end-diastolic dimension Z score > +2.0
  * Biventricular physiology with systemic left ventricle
* Must receive guideline directed heart failure as defined by the American Heart Association, American College of Cardiology, and Heart Failure Society of America 118
* Have been unresponsive or poorly responsive to at least 3 months of maximum guideline directed treatments.

Exclusion Criteria

* Listed for heart transplantation (as UNOS status 1A) or hospitalized while waiting for transplant (while on inotropes or with ventricular assist device)
* Cardiovascular surgery of percutaneous intervention to palliate or correct congenital cardiovascular malformations within 3 months of the screening visit. Patients anticipated to undergo corrective heart surgery during the 12 months after entry into Part 1A/1B.
* Previous heart transplant recipient
* Unoperated primary obstructive or severe regurgitant valve (aortic, pulmonary, or tricuspid) disease, or significant systemic ventricular outflow obstruction or aortic arch obstruction.
* Severe mitral valve disease
* Restrictive or hypertrophic cardiomyopathy
* Cardiogenic shock
* Currently on extracorporeal membrane oxygenation support
* Ventricular assist device support
* Lethal, uncontrollable arrhythmia defined as an arrhythmia resulting in hemodynamic instability requiring need for defibrillation, continuous intravenous anti-arrhythmic medication or mechanical circulatory support
* Patients with persistent atrial fibrillation requiring specific pharmacotherapy
* Amyloidosis
* Ischemic dilated cardiomyopathy
* Clinical history of malignant neoplasm within 5 years (with the exception of curatively treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma)
* Serious neurologic disorder including loss of vision, stroke, or paralysis
* High-grade pulmonary embolism requiring interventional catheter procedure or pulmonary hypertension requiring use of pulmonary vasodilators including phosphodiesterase inhibitor or nitric oxide
* High-grade renal failure [eGFR<45] mL/min/1.73 m2 - serum potassium >5.3 mmol/L
* Multiple organ failure
* Non-cardiac condition that limits life span for <1 year
* Uncontrolled diabetes (HbA1c >9%) at screening
* Active infection (including endocarditis) requiring pharmacotherapy
* Sepsis
* Active hemorrhagic disease (e.g., gastrointestinal bleeding, injury)
* History of cardiac transplantation
* Immune system-altering medications, or immunosuppressive therapy at the time of enrolment or within the prior 12 weeks
* Dystrophin-associated cardiomyopathy confirmed by standard cardiomyopathy panel testing
* Confirmed myocarditis at time of screening
* Elevated LFTs greater than 2 times upper limit of normal at time of consent
* Elevated WBC greater than upper limit of normal as defined by local lab at time of consent
* Presence of HLA antibodies specific for therapeutic study product
* History of noncompliance, alcohol abuse, recreational drug use, or incarceration within the last year
* Currently pregnant or breastfeeding

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with freedom from any Common Toxicity Criteria for Adverse Events (CTCAE) Grade 3 or greater | End of study, around 12 months post-intervention
  Proportion of participants with freedom from any Common Toxicity Criteria for Adverse Events (CTCAE) Grade 3 or greater AE that is probably or related to the IP throughout the duration of the study will be recorded. Results can vary from 0 to 100% and higher proportion correlates with better outcome.
  TCAE Grade 3 is defined as severe or medically significant not immediately life-threatening; hospitalization or prolongation of hospitalization.
  Grade 4 and 5 AEs include composite of: death, life-threatening events, initial or prolonged hospitalization, disability of permanent damage and congenital anomaly/birth defects.
Maximum tolerated dose (MTD) in patients with dilated cardiomyopathy | End of study, around 12 months post-intervention
  If two patients in a dosing group have a related SAE or Dose Limiting Toxicity (DLT), then the previous dosing group will be defined as MTD.

SECONDARY OUTCOMES:
Change of left ventricular ejection fraction (LVEF) from baseline | Baseline, 3-month, 6-month, and 12-month post-intervention
  Change of left ventricular ejection fraction (LVEF) between baseline, 3-month, 6-month, and 12-month follow-up determined by echocardiography and cardiac MRI.
Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) levels from baseline | Baseline, 3-month, 6-month, and 12-month post-intervention
  N-terminal pro b-type natriuretic peptide (NT-proBNP) levels will be collected on infusion days, and all post infusion follow up visits.
Change of 6-minute walk test (6MWT) results | Baseline, 3-month, 6-month, and 12-months post-intervention
  A 6-minute walk test (6MWT) will be completed at baseline, 3-month, 6-month, and 1-year visits to measure functional status if the participant is developmentally appropriate. Distance in meters will be measured until the participant can either walk 6 minutes, or they become too exhausted.
Change in quality-of-life validated survey scores in Peds Quality of Life (QOL) survey | Baseline, 3-month, 6-month and 12-month post-intervention
  Change in quality-of-life validated survey scores in Peds Quality of Life (QOL) survey (≥4 years - < 18 years). Total possible score ranges from 0 to 100 and higher scores indicate better QOL.
Change in Kansas City Cardiomyopathy Questionnaire | Baseline, 3-month, 6-month and 12-month post-intervention
  Change in Kansas City Cardiomyopathy Questionnaire will be recorded (≥18 years - ≤30 years). KCCQ scores are scaled from 0 to 100 and summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.

CONTACTS AND LOCATIONS:
Overall Officials: William Mahle, MD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - Hughes Spalding Children's Hospital, Atlanta, Georgia
  - Egleston Children's Hospital, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Scottish Rite Children's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification and publication.
  Data will be shared with Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, to achieve aims in the approved proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following the publication and then for a minimum of 5 years
Access Criteria: Proposals should be directed to mahlew@kidsheart.com and Edwin.horwitz@emory.edu. To gain access, data requestors will need to sign a data access agreement.